CLINICAL TRIAL: NCT07065799
Title: Respiratory Strategies in COPD Patients With Persistent Hypercapnia Following Exacerbation: A Multicenter, Non-inferiority, Randomized, Crossover Study
Brief Title: Respiratory Strategies in COPD Patients With Persistent Hypercapnia Following Exacerbation
Acronym: RESPHYC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Azienda Sanitaria dell'Alto Adige (Other); Ospedale San Donato (Other); Azienda Unita Sanitaria Locale di Piacenza (Other); Policlinico Universitario, Catania (Other); Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Prof., IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: n° 22/2024/Disp/AOUBo
Record Dates: First submitted 2024-05-17; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: COPD; Hypercapnia; Exacerbation Copd
Keywords: COPD; hypercapnia; NHF; HMV; PaCO2
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, controlled, crossover, non-inferiority
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): NHF/LTOT
  Interventions: Device: Group 1: NHF/LTOT
- Group 2 (Active Comparator): HMV/LTOT
  Interventions: Device: Group 2: HMV/LTOT

INTERVENTIONS:
Device: Group 1: NHF/LTOT — Patients assigned to this group will start NHF (Nasal High Flow) + oxygen therapy at home and undergo a preliminary trial with NHF to set the optimal flow using the MyAIRVO 3 (Fisher & Paykel Healthcare, Auckland, New Zealand) with Optiflow+Duet interface. Patients assigned to this group will be required to use NHF for a minimum of 6 hours per night during sleep, while no restrictions will be set on the duration of use or the times of day to use the device. Patients will continue this treatment for a period of 3 months. At the end of the 3 months, there will be a one-week wash-out period, after which treatment with the control respiratory strategy (HMV+LTOT) will begin.
  Arms: Group 1
Device: Group 2: HMV/LTOT — Patients assigned to this group will start home treatment with HMV (Home Mechanical Ventilation) + oxygen therapy and will be treated with HMV using a pressure support (PS) ventilator. HMV will be administered via nasal mask or full face mask according to patients' preference. Patients assigned to this group will be required to use HMV for a minimum of 6 hours per night in addition to daily home oxygen therapy for at least 15 hours. Moreover, no restrictions will be imposed on the duration of use or the times of day to use the device. Patients will continue this treatment for a period of 3 months. At the end of the 3 months, there will be a one-week wash-out period, after which treatment with the studied respiratory strategy (NHF+LTOT) will begin.
  Arms: Group 2

SUMMARY:
This multicenter, cross-over study aims to investigate the effects of two different respiratory strategies, the use of high flow nasal cannula (NHF) and the use of home mechanic ventilation (HMV), both associated with standard oxygen therapy, in patients with COPD and persistent hypercapnia following a severe acute exacerbation.

The purpose is to evaluate whether the clinical benefits, in terms of reduction in PaCO2 levels, resulting from the use of NHF are non-inferior to those obtained from the use of HMV.

Partecipants will be randomized at 1:1 ratio into two groups:

group 1: will start the respiratory strategy under study (NHF + standard oxygen therapy) as first treatment group 2 will start the control respiratory strategy (HMV + standard oxygen therapy) as first treatment.

The study has a crossover design: each patient will undergo treatment with the two different respiratory strategies, NHF and HMV, each lasting for 3 months

DETAILED DESCRIPTION:
This multicenter, cross-over study aims to investigate the effects of two different respiratory strategies, the use of high flow nasal cannula (NHF) and the use of home mechanic ventilation (HMV) both associated with standard oxygen therapy, in patients with COPD and persistent hypercapnia following a severe acute exacerbation. The purpose of this study is to evaluate whether the clinical benefits, in terms of reduction in PaCO2 levels, resulting from the use of NHF are non-inferior to those obtained from the use of HMV.

Patients will be randomly assigned through a simple randomization list, stratified by recruiting center, generated by the Stata statistical software. Based on this list, patients will be divided into two groups: group 1 will start as the first treatment with the respiratory strategy under study (NHF + standard oxygen therapy) and group 2 will start as the first treatment with the control respiratory strategy (HMV + standard oxygen therapy). Randomization will occur at a 1:1 ratio. The study has a crossover design; each patient will undergo treatment with the two different respiratory strategies, NHF and HMV, each lasting for 3 months. To minimize the carry-over effect, a washout period of 7 days between respiratory supports will be scheduled. Therefore, considering the washout period, the total treatment duration is 25 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acquisition of informed consent form
* Patients with COPD
* Persistent hypercapnia (PaCO2 >53 mmHg) 2-4 weeks after an acute hypercapnic exacerbation of COPD requiring NIV.
* pH value >7.35.
* Chronic hypoxemia (PaO2 <55mmHg or <60mmHg if at least one of the following criteria is present: polycythemia, pulmonary hypertension or Chronic Pulmonary Heart Disease, >30% of sleep time with SpO2 < 90% measured with a pulse oximeter)

Exclusion Criteria:

* BMI >30 kg/m2
* Clinically significant obstructive sleep apnea syndrome (patients in whom there was a clinical suspicion of OSA syndrome based on clinical review or overnight oximetry will go further testing with limited respiratory polygraphy)
* Neuromuscular or chest wall diseases
* Need for intubation and invasive mechanical ventilation during exacerbation
* Use of home non-invasive mechanical ventilation or CPAP
* Contraindications for NIV
* Presence of cognitive impairment that would prevent informed consent into the trial
* Patients with active and unstable coronary artery syndrome
* Patients suffering from malignancies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the non-inferiority of the change in PaCO2 levels measured during treatment with NHF respiratory support compared to HMV respiratory support, both associated with standard oxygen therapy. | T0 (baseline), T1 (+3months), T2 (+6months)
  Unity of measurement: mmHg

SECONDARY OUTCOMES:
Evaluation of the time required for setting up and adjusting the two respiratory strategies. | T0 (baseline), T1 (+3months), T2 (+6months)
  Unit of measurement: days
Evaluation of PaO2 levels measured via arterial blood gas analysis | T0 (baseline), T1 (+3months), T2 (+6months)
  Unit of measurement: mmHg
FVC, FEV1 | T0 (baseline), T1 (+3months), T2 (+6months)
  Measured by spirometry Unit of measurement for FVC and FEV1: L
Evaluation of exercise capacity measured using the 6-minute walk test (6MWT) | T0 (baseline), T1 (+3months), T2 (+6months)
  Unit of measurement: meters
Evaluation of dyspnea measured using the Medical Research Council Dyspnea score | aT0 (baseline), T1 (+3months), T2 (+6months)
  mMRC score ranges from 0 to 4. 0=No dyspnea symptoms 4=severe dyspnea
Evaluation of quality of life measured using the St. George's Respiratory Questionnaire | T0 (baseline), T1 (+3months), T2 (+6months)
  SGRQ's Total Score ranges between 0 and 100, where 0 is maximum quality of life and 100 is lowest quality of life
Evaluation of quality of sleep measured using the Pittsburg Sleep Quality Index | T0 (baseline), T1 (+3months), T2 (+6months)
  PSQI ranges from 0 to 21, higher score indicate worse sleep quality
Evaluation of compliance to respiratory supports measured by downloading usage data from the respiratory support. | T1 (+3months), T2 (+6months)
  Time of usage of the respiratory support in hours/day and hours/night.
Evaluation of tolerance to respiratory supports meauserd using visual analog scales | T1 (+3months), T2 (+6months)
  Visual analog scale ranges between 0 to 10, 0=minimum tolerance 10=maximum tolerance
Evaluation of frequency of exacerbations measured by counting the numbers of exacerbations occurred. | three, six and 12 month since the beginning of the treatment
  Unit of measurement: number of events
Evaluation of severity of exacerbations and subsequent hospitalizations measured by counting the number of exacerbations that required hospitalizations | T1 (+3months), T2 (+6months) and T3 (+12months)
  Unity of measurement: number of exacerbation that required hospitalisation
Evaluation of survival measured by mortality analysis | T1 (+3months), T2 (+6months) and T3 (+12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Pisani, Prof.ssa, Principal Investigator — University of Bologna
Locations (5):
- Italy (5):
  - Ospedale S Donato, Arezzo
  - Bolzano Hospital, Bolzano
  - Azienda Ospedaliera Universitaria Policlinico "G. Rodolico-Sn Marco", Catania
  - ICS Maugeri Spa Società Benefit IRCCS, Pavia
  - Azienda Unità Sanitaria Locale, Piacenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy PB, Rehal S, Arbane G, Bourke S, Calverley PMA, Crook AM, Dowson L, Duffy N, Gibson GJ, Hughes PD, Hurst JR, Lewis KE, Mukherjee R, Nickol A, Oscroft N, Patout M, Pepperell J, Smith I, Stradling JR, Wedzicha JA, Polkey MI, Elliott MW, Hart N. Effect of Home Noninvasive Ventilation With Oxygen Therapy vs Oxygen Therapy Alone on Hospital Readmission or Death After an Acute COPD Exacerbation: A Randomized Clinical Trial. JAMA. 2017 Jun 6;317(21):2177-2186. doi: 10.1001/jama.2017.4451. PMID 28528348
- [Background] Ergan B, Oczkowski S, Rochwerg B, Carlucci A, Chatwin M, Clini E, Elliott M, Gonzalez-Bermejo J, Hart N, Lujan M, Nasilowski J, Nava S, Pepin JL, Pisani L, Storre JH, Wijkstra P, Tonia T, Boyd J, Scala R, Windisch W. European Respiratory Society guidelines on long-term home non-invasive ventilation for management of COPD. Eur Respir J. 2019 Sep 28;54(3):1901003. doi: 10.1183/13993003.01003-2019. Print 2019 Sep. PMID 31467119
- [Background] Oczkowski S, Ergan B, Bos L, Chatwin M, Ferrer M, Gregoretti C, Heunks L, Frat JP, Longhini F, Nava S, Navalesi P, Ozsancak Ugurlu A, Pisani L, Renda T, Thille AW, Winck JC, Windisch W, Tonia T, Boyd J, Sotgiu G, Scala R. ERS clinical practice guidelines: high-flow nasal cannula in acute respiratory failure. Eur Respir J. 2022 Apr 14;59(4):2101574. doi: 10.1183/13993003.01574-2021. Print 2022 Apr. PMID 34649974
- [Background] Storgaard LH, Hockey HU, Laursen BS, Weinreich UM. Long-term effects of oxygen-enriched high-flow nasal cannula treatment in COPD patients with chronic hypoxemic respiratory failure. Int J Chron Obstruct Pulmon Dis. 2018 Apr 16;13:1195-1205. doi: 10.2147/COPD.S159666. eCollection 2018. PMID 29713153
- [Background] Weinreich UM, Juhl KS, Soby Christophersen M, Gundestrup S, Hanifa MA, Jensen K, Andersen FD, Hilberg O, Storgaard LH. The Danish respiratory society guideline for long-term high flow nasal cannula treatment, with or without supplementary oxygen. Eur Clin Respir J. 2023 Feb 23;10(1):2178600. doi: 10.1080/20018525.2023.2178600. eCollection 2023. PMID 36861118
- [Background] Pisani L, Vega ML. Use of Nasal High Flow in Stable COPD: Rationale and Physiology. COPD. 2017 Jun;14(3):346-350. doi: 10.1080/15412555.2017.1315715. Epub 2017 May 1. PMID 28459282